CLINICAL TRIAL: NCT07292025
Title: A Randomized, Double-blind, Active-controlled, Multicenter, Phase 1 Trial to Investigate the Safety and Efficacy of JTM201 in Subjects With Post-stroke Upper Limb Spasticity
Brief Title: Phase 1 Trial of JTM201 in Subjects With Post-stroke Upper Limb Spasticity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jetema Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JTM201-ULP1
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Upper Limb Spasticity Post-Stroke
Keywords: ULP; upper limb spasticity post-stroke
MeSH Terms: interventions — Saline Solution; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JTM201 (Experimental)
  Interventions: Drug: JTM201 in normal saline
- Botox (Active Comparator)
  Interventions: Drug: BOTOX 100U in normal saline

INTERVENTIONS:
Drug: JTM201 in normal saline — Max 360 U of Test drug IM
  Arms: JTM201
Drug: BOTOX 100U in normal saline — Max 360 U of BOTOX IM
  Arms: Botox

SUMMARY:
Phase 1 trial to evaluate the safety and efficacy of JTM201 compared with 'Botox® Inj.' in subjects with post-stroke upper limb spasticity

ELIGIBILITY:
Inclusion Criteria:

* Subjects (or legal representatives) who voluntarily decided the participation of the study and provide written informed consent
* Subjects ≥ 19 years of age, inclusive
* Subjects who was diagnosed stroke at least 6 months prior to screening
* Subjects with MAS score with the wrist flexor score ≥2 and at least one of the elbow flexor or finger flexor score ≥1
* Subjects with a Disability Assessment Scale (DAS) score ≥2 in at least one functional domain, hygiene, dressing, limb position, or pain, selected as the primary treatment goal
* Female subjects who are non-childbearing potential, or childbearing* subjects who are not pregnant, or breastfeeding, a negative serum pregnancy result during screening, and women and men of childbearing potential who agree to use medically acceptable contraceptive methods** or to be sexual abstinence during the study period

Exclusion Criteria:

* Any medical condition that may affect neuromuscular function (eg, myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis)
* Subjects with dysphagia that, in the judgment of the investigator, may interfere with study participation
* Subjects with fixed joint/muscle contracture* at the planned injection sites
* Subjects with severe muscle atrophy at the planned injection sites
* Subjects with skin abnormalities such as infection, skin disease, or scar at the planned injection sites
* History of acute deterioration in pulmonary function within 3 months prior to screening [including but not limited to hospitalization due to asthma or COPD exacerbation, or pneumonia]
* History of chemodenervation using phenol or alcohol, or surgery at the planned injection site within 24 weeks prior to screening, or scheduled for treatment or surgical intervention during the study
* History of tendon lengthening of the study limb within 24 weeks prior to screening, or scheduled surgical intervention at the planned injection site during the study
* Previous treatment with botulinum toxin of any serotype in any area within 24 weeks prior to screening
* Subjects with ongoing treatment with intrathecal Baclofen
* Subjects who require the administration of concomitant medications or implementation of concomitant therapies during the study period

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Modified Ashworth Scale score of Wrist Flexor | Week 4, Week 8, Week 12
  The Modified Ashworth Scale (MAS), a clinical scale used to assess muscle spasticity, was administered with the subject placed in a supine position. The investigator performing the assessment was required to be adequately trained and familiar with the MAS grading criteria, and the same evaluator was used throughout the clinical study whenever possible.
Change from baseline in Modified Ashworth Scale score of Elbow Flexor, Finger Flexor | Week 4, Week 8, Week 12
  The Modified Ashworth Scale (MAS), a clinical scale used to assess muscle spasticity, was administered with the subject placed in a supine position. The investigator performing the assessment was required to be adequately trained and familiar with the MAS grading criteria, and the same evaluator was used throughout the clinical study whenever possible.
Proportion of subjects with at least 1-point improvement from baseline in the Modified Ashworth Scale score for the Wrist Flexor, Elbow Flexor, Finger Flexor | Week 4, Week 8, Week 12
  The Modified Ashworth Scale (MAS), a clinical scale used to assess muscle spasticity, was administered with the subject placed in a supine position. The investigator performing the assessment was required to be adequately trained and familiar with the MAS grading criteria, and the same evaluator was used throughout the clinical study whenever possible.
Changes from baseline in Disability Assessment Scale score | Week 4, Week 8, Week 12
  The Disability Assessment Scale (DAS) was evaluated by the investigator through an interview with the subject. The assessment was performed by the same investigator throughout the clinical study whenever possible to assess Hygiene, Dressing, Limb Position, and Pain.
Global Assessment Scale evaluated by investigator | Week 4, Week 8, Week 12
  The overall improvement in muscle stiffness was assessed using the Global Assessment Scale (GAS) by both the investigator and the subject at Weeks 4, 8, and 12 after administration of the investigational product.
Global Assessment Scale evaluated by patients | Visit 3, 4, 5
  The overall improvement in muscle stiffness was assessed using the Global Assessment Scale (GAS) by both the investigator and the subject at Weeks 4, 8, and 12 after administration of the investigational product.
Change from baseline in Caregiver Burden Scale completed by caregiver | Week 4, Week 8, Week 12
  The Caregiver Burden Scale, a tool used to assess the level of caregiver assistance required for activities of daily living, was evaluated using a 5-point Likert scale for four tasks related to the affected arm (arm with spasticity).

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Boramae Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No